CLINICAL TRIAL: NCT05285761
Title: ECR Visant à évaluer l'Effet d'Une Intervention Sur la Diffusion d'Informations (Conduite de la Diversification Alimentaire) Sur le Comportement de Nourrissage Des Parents, le Comportement Alimentaire et le Statut pondéral de l'Enfant
Brief Title: feediNg gUidelines infanT RandomIzEd coNtrolled Trial
Acronym: NUTRIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Institut de Recherche en Santé Publique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Burgundy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2020-A01941-38
Record Dates: First submitted 2022-03-03; First posted 2022-03-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Complementary feeding; Delivery of information; Recommendations; BMI z-score; Parental feeding practices; Infant eating behavior; Smartphone application; RCT

STUDY DESIGN:
Intervention Model Description: Intervention run between 3 and 36 months of the children, randomisation of children within a control (n=165) or intervention group (n=165).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Parents are informed that the aim of the study concerns the effect of the dissemination of information relating to the conduct of complementary feeding on parental feeding behavior during meals as well as on the eating behavior of their child, but they are blinded to the group (intervention vs. control) to which they are allocated.
  Parents are randomized into 2 groups (intervention vs. control) via the smartphone application. The investigators conduct the study without information on group allocation. The investigators will analyse the data without information on group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paper brochure + smartphone application (Experimental): Parents will receive the paper brochure (new communication support developed by Santé publique France (the French Public Health Agency)), which is the current official information on complementary feeding (CF) in France. They will also receive the new recommendations relating to complementary feeding through an educational device in the form of a smartphone application. This app will deliver information and very short videos illustrating various aspects of responsive feeding during CF and taking up the themes of the paper brochure. These 106 messages will be delivered regularly from the 3rd month until the 36th month of the child. Parents will also receive generic information (48 messages) contained in the health record and in connection with the general development.
  Interventions: Behavioral: Provision of extended information on the conduct of complementary feeding
- paper brochure (Active Comparator): Parents will receive the paper brochure (new communication support developed by Santé publique France (the French Public Health Agency)), which is the current official information on complementary feeding (CF) in France. Parents will also receive generic information (48 messages) contained in the health record and in connection with the general development.
  Interventions: Behavioral: Provision of current official information on complementary feeding

INTERVENTIONS:
Behavioral: Provision of extended information on the conduct of complementary feeding — Parents will receive the paper brochure (new communication support developed by Santé publique France (the French Public Health Agency)), which is the current official information on complementary feeding (CF) in France. Parents will receive generic information contained in the health record and in connection with the general development. These 48 messages will be delivered regularly by a smartphone application from the 3rd months until the 36th months of the child.
  In addition to the paper brochure and the generic information, parents in the intervention group will also receive the new recommendations relating to CF through an educational device (in the form of a smartphone application). This app will deliver information and very short videos illustrating various aspects of responsive feeding during CF and taking up the themes of the paper brochure. These 106 messages will be delivered regularly from the 3rd months until the 36th months of the child.
  Arms: paper brochure + smartphone application
Behavioral: Provision of current official information on complementary feeding — Parents will receive the paper brochure (new communication support developed by Santé publique France (the French Public Health Agency)), which is the current official information on complementary feeding (CF) in France. Parents will also receive generic information contained in the health record and in connection with the general development. These 48 messages will be delivered regularly by a smartphone application from the 3rd months until the 36th months of the child.
  Arms: paper brochure

SUMMARY:
The purpose of this randomized controlled trial is to conduct an intervention aimed at providing first-time parents with information on the conduct of complementary feeding through a paper brochure and a smartphone application, to test the effect of this intervention (compared to usual care, i.e. receiving the paper brochure only), on infant corpulence at 36 and 48 months of age, and parental feeding practices and infant eating behavior up to 36 months of age.

DETAILED DESCRIPTION:
The intervention will consist in the dissemination of new French recommendations relating to complementary feeding, in particular in connection with an educational device in the form of a smartphone application delivering relevant infant feeding messages in due time between the ages of 3 and 36 months.

In France, new recommendations relating to complementary feeding are disseminated to the general public by Santé publique France (the French Public Health Agency) since September 2021 in the form of a paper brochure. Based on the recommendations of this brochure, a smartphone application was developped.

Parents in the intervention (n=165) and control groups (n=165) will receive the paper brochure when the infant will reach the age of 3 months. In the intervention group, a smartphone application will additionnaly support this paper medium, providing information and very short videos illustrating some aspects of responsive feeding during complementary feeding and taking up the themes of the paper brochure. Information will be sent through the smartphone app regularly until the children reach the age of 36 months. In total 106 specific messages will be sent to parents between 3 and 36 months in the intervention group and 48 generic messages to both groups.

The main objective is to determine if the intervention is associated to a difference between the BMI z-score at the age of 36 months of the children of the parents of the intervention group, compared with those of the control group. Parental feeding practices and infant eating behavior will be evaluated several times during the follow-up from the 3rd month of the infant until his 48th month with various validated questionnaires from the literature (n=330) and with behavioral evaluations (n=130, 65 in each group) carried out during meals filmed in the laboratory and at the participants' homes.

Our goal is to involve a total of 330 parents and children (with only first-time parents); the first 30 children will allow us to test the device but their data may not be included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* first-time parents
* child age is between 1 and 54 days
* parents living in Dijon and its surroundings (~ 70 km around Dijon)
* parents who master enough the french language to understand and answer self-reported questionnaires

Exclusion Criteria:

* no affiliation to a social security scheme
* parents of a child born before 31 weeks of amenorrhea
* parents of a child presenting since birth with pathologies likely to have a strong impact on his diet or his feeding habits (allergy to cow's milk proteins, feeding through a nasogastric tube or gastrostomy, congenital defect of the digestive tract, oral feeding disorders)
* parents of a child with a multiple pregnancy (≥ 3 children).
* in the event of a twin birth, the follow-up for this study only focuses on one of the children (according to a random draw)
* additional exclusion criteria for participation in filmed meals from the age of 11 months: children with food allergies or intolerances or suffering from celiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Body mass index z-score at the age of 36 months | End of intervention (at the age of 36 months)
  Z-score of the body mass index (BMI, kg / m²) at the age of 36 months of the child of the parents included in the study, calculated from measurements of the child's weight and height at the age of 36 months (carried out in the laboratory) and according to the WHO references.

SECONDARY OUTCOMES:
Body mass index z-score at the age of 48 months | Follow-up (at the age of 48 months)
  Z-score of the body mass index (BMI, kg / m²), calculated from measurements of the child's weight and height at the age of 48 months (parent-reports of the measurements contained in the child health record) and according to the WHO references.
Children's eating behaviour (self-reported by parents) | at the ages of 12 and 36 months
  Parent-reports using the french version of the Child Eating Behaviour Questionnaire adapted for toddlers (CEBQ-T) which is a validated questionnaire. The questionnaire is composed of 31 items. Parent answers to each item using a 6-category scale (never, rarely, sometimes, often, always, I don't know). The items are then grouped to define 7 dimensions : 'food responsiveness', 'enjoyment of food', 'satiety responsiveness', 'food fussiness', 'slowness in eating', 'emotional overeating', and 'external food cue responsiveness'. Higher scores mean higher behaviours.
Infant appetite control abilities (self-reported by parents) | at the ages of 12 and 36 months
  Parent-reports at the ages of 12 and 36 months using a validated questionnaire. Parent answers to 9 items, which are then grouped to define 2 dimensions: 'Caloric compensation' and 'Eating in the absence of hunger' (EAH). Parent answers to items using a 5-category scale (never, rarely, sometimes, often, always). Higher scores mean higher behaviours.
Infant appetite control abilities (behavioral observation) | at the age of 11 months
  Infant caloric compensation ability during 2 meals at the laboratory at the age of 11 months (calculation of "COMPX" scores)
Infant appetite control abilities (behavioral observation) | at the age of 30 months
  Infant Eating in the Absence of Hunger (EAH) during a meal at the laboratory at the age of 30 months (assessment of quantities and choice of food consumed during 10 minutes after a meal, i.e. when the child is no longer hungry).
Parental feeding practices (self-reported by parents) | at the ages of 12, 24, 36 months
  Parent-reports at the ages of 12, 24, 36 months using the validated French version of the Child Feeding Practices Questionnaire. Parent answers to items 1-12 using a 6-category scale (never, rarely, sometimes, often, always, not concerned). Parent answers to items 13-39 using a 5-category scale (not at all true, bit true, moderately true, rather true, very true). The 39 items are grouped to define 10 dimensions: 'Monitoring' , 'Child control' , 'Emotion Regulation' 'Positive habits', 'Restriction for weight control', 'Restriction for health reasons', 'Food as reward', 'Teaching nutrition', 'Modeling' , 'Responsibility'. Higher scores mean higher behaviors.
Parental feeding practices (behavioral observation) | at the ages of 32 and 36 months
  Filmed meal at the laboratory at the age of 36 months to observe parental strategies for coping with food refusal (parents will choose from a selection a vegetable that is not appreciated by the child. The strategies the parent will use to get the food tasted will be recorded.)
  + Filmed meal at participants' home at the age of 32 months in order to assess the quality of interactions in a more natural context.
  The overall behaviors of the infant during the meal (e.g.: "turns his head", "signals with his hand that he is no longer hungry", etc.) as well as the behaviors of the parent who feeds (e.g.: "talks to encourage her infant", "takes a break from feeding", "flys the plane with the spoon", etc.) will be described on the basis of a video analysis thanks to the establishment of ethograms.
Introduction of complementary foods | at the ages of 3, 6, 12, 18, 24, 36, 48 months
  Parent-reports using a questionnaire from a previous research (RCT ECAIL). This questionnaire is composed of 93 items relating to breastfeeding (age of stopping and reasons), milks (type of milks offered to the baby), age and reasons for starting complementary feeding (CF) and items representing different drinks and complementary foods. Parent answers to each food item using a 5-category scale (not yet introduced, only once, 2 or 3 times, more often, every day or almost every day) (higher scores mean higher consumption frequency) and indicates the age of introduction as soon as the consumption frequency is higher than 'only once'.
  Particular interest will be given to : 'age at the start of CF', 'reasons for starting CF', 'diversity of foods introduced between 4 and 6 months', 'diversity of major allergens introduced between 4 and 6 months', 'consumption frequency' and 'age of introduction' of various food groups.
Food frequency and food acceptance | at the age of 36 months
  Parent-reports using a questionnaire from a previous research (ANR OPALINE). This questionnaire is composed of 257 food items. Parent answers to each item using a 5-category scale (almost every day, 1 to 3 times a week, 1 to 3 times per month, less than once a month, never) to assess frequency (higher scores mean higher consumption frequency) and using a 4-point scale (++, +, -, --) to assess liking (higher scores mean higher liking).
Food texture exposure and acceptance | at the age of 12 months
  Parent-reports using a summarized version of a questionnaire developed to characterize the pattern of food texture exposure in French children aged 4-36 months. This questionnaire is composed of items representing foods commonly used in France in different texture combinations (puree, pieces, raw, cooked, etc.)). Parent answers to each item using a 4-category scale (not offered, spit out, eaten with difficulty, eaten without difficulty). Higher scores mean higher behaviors.
Child feeding skills | at the ages of 12 and 36 months
  Parents will report children general feeding skills (holding a spoon in the mouth alone, eating with fingers, self-feeding with a fork, etc.) on a 5-category scale (often, sometimes, rarely, never, I don't know). Higher scores mean higher feeding skills.
Meal context - FPSQ | at the ages of 12, 24, 36 months
  Parent-reports at the ages of 12, 24, 36 months using translated extracts from the validated Feeding Practices and Structure Questionnaire. Parent answers to 7 items using a 5-category scale (never, rarely, sometimes, often, always). Items are grouped to define 3 dimensions : 'Family meal setting', ' Structured Meal Timing', 'Structured Meal Setting '. Higher scores mean higher behaviours.
Meal context - FFBS | at the ages of 12, 24, 36 months
  Parent-reports at the ages of 12, 24, 36 months using translated extracts from the validated Family Food Behavior Survey. Parent answers to 12 items using a 5-category scale (never true, rarely true, sometimes true, often true, always true). Items are grouped to define 2 dimensions : 'Maternal control' and 'Organization of eating environment'. Higher scores mean higher behaviours.
Maternal distractions during feeding - Use of technological distractors | at the ages of 12, 24, 36 months
  Parent-reports at the ages of 12, 24, 36 months using an adapted version of the Maternal Distraction Questionnaire which is a validated questionnaire. Higher scores mean higher behaviour.
Maternal distractions during feeding - Perceived Distraction | at the ages of 12, 24, 36 months
  Parent-reports at the ages of 12, 24, 36 months using an adapted version of the Maternal Distraction Questionnaire which is a validated questionnaire. Higher scores mean higher perception
Knowledge about infant nutrition | at the age of 36 months
  Parent-reports using a questionnaire developped by De Rosso et al. (in press). This questionnaire is composed of 30 items representing various infant feeding recommendations. Parent first answers to each item on a dichotomous true/false scale and then indicates how sure he/she is of his/her answer on a 4-category scale (I am not at all sure, I am rather unsure, I am rather sure, I am completely sure). Two dimensions are assessed : Knowledge accuracy and Knowledge certainty.Higher scores mean higher accuracy/certainty.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Schwartz, PhD, Principal Investigator — INRAE UMR CSGA
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: March 2025
Access Criteria: Public
URL: https://osf.io/

REFERENCES:
- [Background] Asta K, Miller AL, Retzloff L, Rosenblum K, Kaciroti NA, Lumeng JC. Eating in the Absence of Hunger and Weight Gain in Low-income Toddlers. Pediatrics. 2016 May;137(5):e20153786. doi: 10.1542/peds.2015-3786. Epub 2016 Apr 18. PMID 27244808
- [Background] Brugailleres P, Chabanet C, Issanchou S, Schwartz C. Caloric compensation ability around the age of 1 year: Interplay with the caregiver-infant mealtime interaction and infant appetitive traits. Appetite. 2019 Nov 1;142:104382. doi: 10.1016/j.appet.2019.104382. Epub 2019 Jul 23. PMID 31348973
- [Background] Brugailleres P, Issanchou S, Nicklaus S, Chabanet C, Schwartz C. Caloric compensation in infants: developmental changes around the age of 1 year and associations with anthropometric measurements up to 2 years. Am J Clin Nutr. 2019 May 1;109(5):1344-1352. doi: 10.1093/ajcn/nqy357. PMID 30997507
- [Background] de Lauzon-Guillain B, Musher-Eizenman D, Leporc E, Holub S, Charles MA. Parental feeding practices in the United States and in France: relationships with child's characteristics and parent's eating behavior. J Am Diet Assoc. 2009 Jun;109(6):1064-9. doi: 10.1016/j.jada.2009.03.008. PMID 19465189
- [Background] Jansen E, Williams KE, Mallan KM, Nicholson JM, Daniels LA. The Feeding Practices and Structure Questionnaire (FPSQ-28): A parsimonious version validated for longitudinal use from 2 to 5 years. Appetite. 2016 May 1;100:172-80. doi: 10.1016/j.appet.2016.02.031. Epub 2016 Feb 18. PMID 26911263
- [Background] McCurdy K, Gorman KS. Measuring family food environments in diverse families with young children. Appetite. 2010 Jun;54(3):615-8. doi: 10.1016/j.appet.2010.03.004. Epub 2010 Mar 20. PMID 20227449
- [Background] Monnery-Patris S, Rigal N, Peteuil A, Chabanet C, Issanchou S. Development of a new questionnaire to assess the links between children's self-regulation of eating and related parental feeding practices. Appetite. 2019 Jul 1;138:174-183. doi: 10.1016/j.appet.2019.03.029. Epub 2019 Mar 26. PMID 30926418
- [Background] Musher-Eizenman D, Holub S. Comprehensive Feeding Practices Questionnaire: validation of a new measure of parental feeding practices. J Pediatr Psychol. 2007 Sep;32(8):960-72. doi: 10.1093/jpepsy/jsm037. Epub 2007 May 28. PMID 17535817
- [Background] Sall NS, Begin F, Dupuis JB, Bourque J, Menasria L, Main B, Vong L, Hun V, Raminashvili D, Chea C, Chiasson L, Blaney S. A measurement scale to assess responsive feeding among Cambodian young children. Matern Child Nutr. 2020 Jul;16(3):e12956. doi: 10.1111/mcn.12956. Epub 2020 Jan 30. PMID 31999399
- [Background] Tournier C, Demonteil L, Ksiazek E, Marduel A, Weenen H, Nicklaus S. Factors Associated With Food Texture Acceptance in 4- to 36-Month-Old French Children: Findings From a Survey Study. Front Nutr. 2021 Feb 1;7:616484. doi: 10.3389/fnut.2020.616484. eCollection 2020. PMID 33598476
- [Background] van der Veek SMC, de Graaf C, de Vries JHM, Jager G, Vereijken CMJL, Weenen H, van Winden N, van Vliet MS, Schultink JM, de Wild VWT, Janssen S, Mesman J. Baby's first bites: a randomized controlled trial to assess the effects of vegetable-exposure and sensitive feeding on vegetable acceptance, eating behavior and weight gain in infants and toddlers. BMC Pediatr. 2019 Aug 1;19(1):266. doi: 10.1186/s12887-019-1627-z. PMID 31370830
- [Background] Ventura AK, Hupp M, Alvarez Gutierrez S, Almeida R. Development and validation of the Maternal Distraction Questionnaire. Heliyon. 2020 Feb 1;6(2):e03276. doi: 10.1016/j.heliyon.2020.e03276. eCollection 2020 Feb. PMID 32025583
- [Derived] Riera-Navarro C, Schwartz C, Ducrot P, Noirot L, Delamaire C, Sales-Wuillemin E, Semama DS, Lioret S, Nicklaus S. A web-based and mobile randomised controlled trial providing complementary feeding guidelines to first-time parents in France to promote responsive parental feeding practices, healthy children's eating behaviour and optimal body mass index: the NutrienT trial study protocol. BMC Public Health. 2024 Sep 27;24(1):2649. doi: 10.1186/s12889-024-20057-z. PMID 39334106